CLINICAL TRIAL: NCT06961656
Title: The Effect of Wound Care Education Using the Jigsaw IV Learning Technique on Nursing Students' Knowledge, Collaborative Learning, and Academic Motivation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Agri Ibrahim Cecen University (Other)
Responsible Party: Principal Investigator, Tugce Kabak Solak, Principal Investigator, Agri Ibrahim Cecen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: AGRSABFTKS001
Record Dates: First submitted 2025-04-19; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Nursing Students; Nursing Education; Jigsaw Technique; Wound Care
Keywords: Jigsaw IV; Nursing students; Wound care; Collaboration; Motivation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wound care training with the Jigsaw IV technique method (Other)
  Interventions: Other: Intervention Group-Jigsaw IV technique
- Wound care training with traditional methods (Other)
  Interventions: Other: Control Group-Traditional methods

INTERVENTIONS:
Other: Intervention Group-Jigsaw IV technique — Wound care training with the Jigsaw IV technique method
  Arms: Wound care training with the Jigsaw IV technique method
Other: Control Group-Traditional methods — Wound care training with traditional methods
  Arms: Wound care training with traditional methods

SUMMARY:
This study aims to investigate the effects of wound care education given with the jigsaw IV learning technique on the knowledge, collaborative learning and motivation levels of nursing students. Second-year nursing students will be divided into two groups with simple randomization. The intervention group will be given a wound care training program with the jigsaw IV technique. The control group will be given wound care training with traditional education. Pre-test data will be collected before the training and post-test data will be collected after the training.

ELIGIBILITY:
Inclusion Criteria:

* Not having taken a wound care education before
* Willing to participate in the study voluntarily

Exclusion Criteria:

* Being a nurse who graduated from secondary school and working in the clinic,
* Having previously established an associate degree program related to health,
* Not participating in theoretical lessons, demonstrations and group work, - The student wants to withdraw from the research at any stage,
* Not filling out the data collection forms or filling them incompletely.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-28 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in Wound Care Knowledge Score | At Baseline, immediately after the training intervention
  The participants' knowledge about wound care will be assessed using a pre-designed knowledge test that measures essential topics such as wound assessment, infection control, dressing types, and aseptic techniques. The knowledge test will be administered immediately before and after the educational interventions. The change in scores will indicate the effectiveness of the training methods.

SECONDARY OUTCOMES:
Change in Collaborative Learning Level | At Baseline, immediately after the training intervention
  The Collaborative Learning Scale will be used to measure students' ability to work in teams, engage in peer discussions, and share knowledge. This scale consists of Likert-type items assessing group interactions, peer collaboration, and group responsibility. A higher scale score indicates a higher level of cooperative learning. The scale will be administered immediately before and immediately after the training intervention.
Change in Academic Motivation Level | At Baseline, immediately after the training intervention
  Academic motivation will be assessed using the Academic Motivation Scale. This scale measures intrinsic and extrinsic motivation factors. A higher scale score indicates a higher level of academic motivation. The academic motivation scale will be administered immediately before and immediately after the training intervention.

IPD SHARING:
Plan to Share IPD: No